CLINICAL TRIAL: NCT06170385
Title: Pediatric Early Rehabilitation in ACute Lymphoblastic LEukemia (PEACE): A Feasibility Study of a Hybrid Delivery Format
Brief Title: Pediatric Early Rehabilitation in Acute Lymphoblastic Leukemia
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-23-0294
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms; Pediatric Cancer; Physical Therapy; Telemedicine
MeSH Terms: conditions — Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Quasi-experimental single group before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Children will participate in six PT sessions over the course of 12 weeks and will be provided with the option to choose their preferred mode of the delivery (i.e., 1:1 in-person, 1:1 virtual, group virtual, or a combination of all). The program will be tailored to the child's age, presenting symptoms, and preferred activities.
  Children and parents/ caregivers will be encouraged to carry out additional tailored PT sessions through their preferred mode of delivery and to access the exercise videos provided in the additional resources section of the HEAL-ME platform.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — Each physical therapy session will commence with a 5-minute warm-up, with fun activities to mobilize the joints and activate the muscles, using the videos available in the HEAL-ME platform. The warm-up session will be followed by a 20 to 40-min program with tailored activities and games comprising jumping, squatting, skipping, balancing, and jogging. The session will finish with a 5-minute cool down with stretching exercises and a relaxation video from the HEAL-ME platform.

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of a hybrid in-person and virtual individualized physiotherapy program using the Healthy Eating and Active Living (HEAL-ME) online platform for children diagnosed with acute lymphoblastic leukemia. We would like to know if this type of hybrid program delivery model is feasible, and if children and their parents are willing and able to participate in the program. We will do this by recording how many, and what type of physiotherapy sessions (in-person or virtual) are completed, what resources offered on the platform are accessed, and how many children complete the assessments.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia is the most common childhood cancer, representing approximately 25% of cancers in children. Improvements in survival rates have resulted in an increased number of children living with neuromuscular and musculoskeletal side effects of cancer treatments-effects that may persist or worsen over the long-term into adulthood.

The overall goal of the study is to determine the feasibility of a tailored physiotherapy (PT) program using an online platform for children diagnosed with acute lymphoblastic leukemia.

A quasi-experimental, single group, before and after intervention feasibility study will be conducted, comprising a convenience sample of a minimum of 10 children between 4 and 17 years of age undergoing or having completed chemotherapy treatment for acute lymphoblastic leukemia. Children will participate in a hybrid 12-week PT program delivered in-person at the Stollery Children's Hospital with educational components provided virtually via the Healthy Eating and Active Living web-based platform. Children will participate in six physical therapy sessions over a period of three months and will have the option to choose the mode of delivery: 1:1 in-person, 1:1 virtual, group virtual, or combination of all. The main outcome will be feasibility, as determined by recruitment and retention rates, completion rates of measurements, adherence to sessions, and safety and acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with acute lymphoblastic leukemia aged between 4 and 17 years (at time of diagnosis) and their mother, father, or primary carer;
2. Undergoing or completed cancer treatment as established by the Children's Oncology Group;
3. Access to the internet through a home computer or tablet;
4. Patient or caregiver is able to speak and comprehend English; and
5. The child is approved by their Oncologist to participate in the program.

Exclusion Criteria:

1. Children with a history of a neurodevelopmental or genetic disorder (i.e., Down syndrome, autism, seizure disorder) prior to the cancer diagnosis; and
2. Children with a concurrent condition (illness, disease, psychiatric disorder), as determined by oncologist or physiotherapist, that would compromise study participation or interpretation of study results.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Retention rate | Post-intervention: 12 weeks
  The number of participants completing the intervention and assessments

SECONDARY OUTCOMES:
Recruitment rate | One year
  Number eligible divided by the number of participants enrolling in the study
Adherence to study intervention | Post-intervention: 12 weeks
  Attendance rates for in-person and virtual physical therapy sessions
Adverse events | One year
  Number of serious and non-serious adverse events
Acceptability | Post-intervention: 12 weeks
  Satisfaction survey
Health-related Quality of Life | Post-intervention: 12 weeks
  Pediatric Quality of Life Inventory Version 4: Total scale score, with higher scores reflecting better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited on the University of Alberta's dataverse
Supporting Information: Study Protocol, ICF, CSR
Time Frame: when the study has been completed and after the findings are published
Access Criteria: Open access